CLINICAL TRIAL: NCT00892710
Title: Randomized Phase II Trial of Pemetrexed vs. Pemetrexed/Bevacizumab vs. Pemetrexed/Carboplatin/Bevacizumab in Patients With Stage IIIB/IV Non-Small-Cell Lung Cancer and ECOG Performance Status 2
Brief Title: Trial of Poor Performance Status Patients (ToPPS)
Acronym: ToPPS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 196
Record Dates: First submitted 2009-04-30; First posted 2009-05-04 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non small cell lung cancer; NSCLC; Pemetrexed; Bevacizumab; Avastin; Carboplatin; Stage IIIB/IV
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pemetrexed/Bevacizumab (Experimental): * Pemetrexed 500 mg/m2 IV given over 10 minutes every 21 days
  * Bevacizumab 15 mg/kg IV every 21 days
  Interventions: Drug: Pemetrexed; Drug: Bevacizumab
- Pemetrexed/Bevacizumab/Carboplatin (Experimental): * Pemetrexed 500 mg/m2 IV given over 10 minutes every 21 days
  * Bevacizumab 15 mg/kg IV every 21 days
  * Carboplatin AUC=5 IV every 21 days
  Interventions: Drug: Pemetrexed; Drug: Bevacizumab; Drug: Carboplatin
- Pemetrexed (Experimental): Pemetrexed 500 mg/m2 IV given over 10 minutes every 21 days
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — 500 mg/m2 IV given over 10 minutes every 21 days
  Other Names: Alimta
Drug: Bevacizumab — 15 mg/kg IV every 21 days
  Other Names: Avastin
  Arms: Pemetrexed/Bevacizumab; Pemetrexed/Bevacizumab/Carboplatin
Drug: Carboplatin — AUC=5 IV every 21 days
  Other Names: Paraplatin
  Arms: Pemetrexed/Bevacizumab/Carboplatin

SUMMARY:
The purpose of this trial is to evaluate three treatment regimens in patients with stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC) with a performance status of 2 and who were not previously treated.

DETAILED DESCRIPTION:
This randomized, Phase II trial will evaluate three treatment regimens in patients with previously untreated stage IIIB/IV Non-Small Cell Lung Cancer (NSCLC) and a performance status (PS) of 2. Patients will be randomized to either pemetrexed alone, pemetrexed and bevacizumab, or pemetrexed, carboplatin, and bevacizumab in a 1:1:1 fashion. All 3 regimens should be tolerable in poor performance status patients with advanced NSCLC. The 3-drug regimen (pemetrexed/carboplatin/bevacizumab) has been modified by lowering the dose of carboplatin, in order to minimize myelosuppression. This trial will be conducted at multiple study sites.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be >=18 years of age.
2. Non-squamous NSCLC (adenocarcinoma or large cell carcinoma). Mixed tumors with small cell anaplastic elements are not eligible. Mixed tumors with squamous histology are acceptable as long as the squamous element is not the dominant histology.
3. Unresectable stage IIIB or stage IV disease. Stage IIIB disease should be ineligible for combined modality therapy (i.e., pleural effusions, pericardial effusions).
4. ECOG performance status of 2.
5. No prior systemic therapy for stage IIIB or stage IV lung cancer.
6. Life expectancy of at least 12 weeks.
7. Patients must have measurable disease per RECIST version 1.1 (see Section 8).
8. Laboratory values as follows:

   * Absolute neutrophil count (ANC) ≥1500/μL
   * Hemoglobin (Hgb) ≥10 g/dL
   * Platelets ≥100,000/μL (≤7 days prior to treatment)
   * AST or ALT and alkaline phosphatase (ALP) must be <2.5 x ULN, or <5 x ULN in patients with liver metastases.
   * Total bilirubin <1.5 x the institutional ULN
   * Calculated creatinine clearance ≥45 mL/min
9. The ability to take folic acid, Vitamin B12, and dexamethasone according to protocol.
10. Women of childbearing potential must have a negative serum or urine pregnancy test performed within 7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
11. Patient must be accessible for treatment and follow-up.
12. Patients must be able to understand the investigational nature of this study and give written informed consent prior to study entry.

Exclusion Criteria:

1. Squamous cell histology. Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient will be ineligible; sputum cytology alone is unacceptable.
2. Patients with active brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if there is no evidence of central nervous system (CNS) disease progression, and at least 2 weeks have elapsed since treatment. Ideally, patients should not still require use of seizure medication or steroids.
3. Patients who have had major surgical procedure (not including mediastinoscopy), open biopsy, or significant traumatic injury within 4 weeks of beginning treatment; or, the anticipation of the need for major surgical procedure during the course of the study.
4. Women who are pregnant or lactating.
5. Minor surgical procedures (with the exception of the placement of portacath or other central venous access) must be completed at least 7 days prior to beginning protocol treatment.
6. History of hypersensitivity to active or inactive excipients of any component of treatment (pemetrexed, bevacizumab, and/or carboplatin).
7. Pulmonary carcinoid tumors.
8. Patients with proteinuria at screening as demonstrated by either:

   * urine protein creatinine (UPC) ratio ≥1.0 at screening OR
   * urine dipstick for proteinuria ≥2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection, and must demonstrate ≤1 g of protein/24 hours to be eligible) (see Appendix B)
9. Patients with a serious non healing wound, active ulcer, or untreated bone fracture.
10. Patients with evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
11. Patients with history of hematemesis or hemoptysis (defined as having bright red blood of ½ teaspoon or more per episode) within 1 month prior to study enrollment.
12. History of myocardial infarction or unstable angina within 6 months of beginning treatment.
13. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and /or diastolic blood pressure >100 mmHg while on antihypertensive medications).
14. New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF) (see Appendix C).
15. Serious cardiac arrhythmia requiring medication.
16. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair, or recent peripheral arterial thrombosis) within 6 months prior to Day 1 of treatment.
17. History of stroke or transient ischemic attack ≤ 6 months prior to beginning treatment.
18. Any prior history of hypertensive crisis or hypertensive encephalopathy.
19. History of abdominal fistula or gastrointestinal perforation ≤ 6 months prior to Day 1 of beginning treatment.
20. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
21. Mental condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
22. Use of any non-approved or investigational agent ≤ 30 days of administration of the first dose of study drug. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.
23. Past or current history of neoplasm other than the entry diagnosis with the exception of treated non-melanoma skin cancer or carcinoma in situ of the cervix, or other cancers cured by local therapy alone and a DFS ≥5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2009-06; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (27):
- United States (27):
  - Mayo Clinic - AZ, Scottsdale, Arizona
  - Genesis Cancer Center, Hot Springs, Arkansas
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Wilshire Oncology Medical Group, LaVerne, California
  - Aventura Medical Center, Aventura, Florida
  - Collaborative Research Group/ Palm Beach Ins of Hem Onc, Boynton Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Regional Cancer Center, Hollywood, Florida
  - Watson Clinic Center for Cancer Care and Research, Lakeland, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - University of Chicago, Chicago, Illinois
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - RHHP/ Hope Cancer Center, Terra Haute, Indiana
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - Toledo Community Oncology Program, Toledo, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Family Cancer Center, Memphis, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Virginia Cancer Institute, Richmond, Virginia

REFERENCES:
- [Derived] Gijtenbeek RG, de Jong K, Venmans BJ, van Vollenhoven FH, Ten Brinke A, Van der Wekken AJ, van Geffen WH. Best first-line therapy for people with advanced non-small cell lung cancer, performance status 2 without a targetable mutation or with an unknown mutation status. Cochrane Database Syst Rev. 2023 Jul 7;7(7):CD013382. doi: 10.1002/14651858.CD013382.pub2. PMID 37419867

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 patients were enrolled/randomized, but never treated due to their reqeust, physician's request or if they were deemed ineligible. 4 of these patients were on the Pemetrexed/Bevacizumab arm and 6 were on the Pemetrexed/Bevacizumab/Carboplatin arm
Period: Overall Study
Arm/Group | Pemetrexed | Pemetrexed/Bevacizumab | Pemetrexed/Bevacizumab/Carboplatin
Started | 48 | 59 | 55
Completed | 0 (Patients remained on study until disease progression or intolerable toxicity occurred) | 0 (Patients remained on study until disease progression or intolerable toxicity occurred) | 0 (Patients remained on study until disease progression or intolerable toxicity occurred)
Not Completed | 48 | 59 | 55

BASELINE CHARACTERISTICS:
Population: Includes all patients who were enrolled (whether they recieved treatment or not)
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed | Pemetrexed/Bevacizumab | Pemetrexed/Bevacizumab/Carboplatin | Total
Number analyzed (Participants) | 48 | 63 | 61 | 172
Age, Continuous [Median (Full Range); unit: years] | 72 [51 to 84] | 72 [50 to 90] | 73 [48 to 90] | 72 [48 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 27 | 72
  Male | 30 | 36 | 34 | 100
Region of Enrollment [Number; unit: participants]
  United States | 48 | 63 | 61 | 172

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 18 months
Population: Includes all enrolled patients whether they recieved treatment or not
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed | Pemetrexed/Bevacizumab | Pemetrexed/Bevacizumab/Carboplatin
Number analyzed (Participants) | 48 | 63 | 61
months | 2.8 [1.5 to 4.1] | 4.0 [2.6 to 6.0] | 4.8 [3.1 to 6.5]

2. Secondary Outcome: Overall Response Rate (ORR), the Number of Patients Who Experience an Objective Benefit From Treatment
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Population: Includes all treated patients
Measure: Number; unit: participants
Arm/Group | Pemetrexed | Pemetrexed/Bevacizumab | Pemetrexed/Bevacizumab/Carboplatin
Number analyzed (Participants) | 48 | 59 | 55
participants | 7 | 18 | 24

3. Secondary Outcome: Time to Progression (TTP)
Description: The Length of Time, in Months, That Patients Remain Alive From Their First Date of Protocol Treatment Until Worsening of Their Disease. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 18 months
Population: Includes all treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed | Pemetrexed/Bevacizumab | Pemetrexed/Bevacizumab/Carboplatin
Number analyzed (Participants) | 48 | 59 | 55
months | 3.5 [1.6 to 5.5] | 5.3 [3.1 to 6.8] | 5.7 [3.8 to 7.1]

4. Secondary Outcome: Time to Treatment Failure (TTTF)
Description: Defined as the Length of Time, in Months, that Patients were Alive from the Date of First Treatment Until Treatment Discontinuation for Any Reason.
Time Frame: 18 months
Population: Includes all treated patients
Measure: Median (Full Range); unit: months
Arm/Group | Pemetrexed | Pemetrexed/Bevacizumab | Pemetrexed/Bevacizumab/Carboplatin
Number analyzed (Participants) | 48 | 59 | 55
months | 2.4 [.5 to 21.2] | 3.1 [.03 to 18.8] | 3.3 [0.2 to 16.1]

5. Secondary Outcome: Overall Survival (OS)
Description: The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 18 months
Population: Includes all enrolled patients, whether or not they were treated
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed | Pemetrexed/Bevacizumab | Pemetrexed/Bevacizumab/Carboplatin
Number analyzed (Participants) | 48 | 63 | 61
months | 7.7 [3.0 to 11.2] | 8.6 [5.3 to 11.2] | 8.7 [5.4 to 13]

6. Secondary Outcome: 6-month and 12-month Overall Survival Probability
Description: Overall Survival = The Length of Time, in Months, That Patients Were Alive From Their First Date of Protocol Treatment Until Death
Time Frame: 12 months
Population: Includes all enrolled patients, whether or not they received treatment
Measure: Number (95% Confidence Interval); unit: probability out of 1
Arm/Group | Pemetrexed | Pemetrexed/Bevacizumab | Pemetrexed/Bevacizumab/Carboplatin
Number analyzed (Participants) | 48 | 63 | 61
probability out of 1
  6-month OS probability | 0.52 [0.37 to 0.65] | 0.61 [0.47 to 0.72] | 0.57 [0.43 to 0.69]
  12-month OS probability | 0.3 [0.18 to 0.43] | 0.32 [0.21 to 0.45] | 0.44 [0.31 to 0.57]

ADVERSE EVENTS:
Time Frame: 18 Months
Arm/Group | Pemetrexed | Pemetrexed/Bevacizumab | Pemetrexed/Bevacizumab/Carboplatin
Serious Adverse Events (participants affected / at risk) | 30/48 | 28/63 | 33/61
Other Adverse Events (participants affected / at risk) | 48/48 | 62/63 | 60/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed (N=48) | Pemetrexed/Bevacizumab (N=63) | Pemetrexed/Bevacizumab/Carboplatin (N=61)
Infections and infestations - Other, pneumonia (Infections and infestations) | 8 | 5 | 4
General disorders and administration site conditions - Other, disease progression (General disorders) | 4 | 4 | 2
Respiratory, thoracic and mediastinal disorders - Other, COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 5
Thromboembolic event (Vascular disorders) | 2 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 2 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Skin infection (Infections and infestations) | 4 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Fever (General disorders) | 2 | 0 | 1
Psychiatric disorders - Other, change in mental status (Psychiatric disorders) | 1 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 2
Investigations - Other, pancytopenia (Investigations) | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Renal and urinary disorders - Other, renal failure (Renal and urinary disorders) | 2 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 1
Stroke (Nervous system disorders) | 0 | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Death NOS (General disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Eye disorders - Other, blindness (Eye disorders) | 1 | 0 | 0
Eye infection (Eye disorders) | 0 | 1 | 0
Gastrointestinal disorders - Other, rectal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorders - Other, small bowel obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, unspecified ulcer (Gastrointestinal disorders) | 0 | 1 | 0
General disorders and administration site conditions - Other, failure to thrive (General disorders) | 0 | 1 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1
Hemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Infections and infestations - Other, intestinal clostridium (Infections and infestations) | 1 | 0 | 0
Infections and infestations - Other, s. maltophilia bacteremia (Infections and infestations) | 0 | 0 | 1
Infections and infestations - Other, Staphylococcus Hominis Bacteremia (Infections and infestations) | 0 | 1 | 0
Investigations - Other, transaminitis (Investigations) | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, acute respiratory insufficiency (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Transient ischemic attacks (Nervous system disorders) | 0 | 0 | 1
Vascular disorders - Other, superior vena cava stenosis (Vascular disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Infections and infestations - Other, gastroenteritis (Infections and infestations) | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed (N=48) | Pemetrexed/Bevacizumab (N=63) | Pemetrexed/Bevacizumab/Carboplatin (N=61)
Fatigue (General disorders) | 29 | 39 | 36
Nausea (Gastrointestinal disorders) | 19 | 23 | 29
Anemia (Blood and lymphatic system disorders) | 18 | 18 | 25
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 26 | 19
Constipation (Gastrointestinal disorders) | 12 | 24 | 21
Anorexia (Metabolism and nutrition disorders) | 15 | 26 | 14
Platelet Count Decreased (Investigations) | 12 | 10 | 24
Neutrophil Count Decreased (Investigations) | 7 | 13 | 21
Edema (General disorders) | 11 | 13 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 16 | 16
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 8 | 14 | 15
Dehydration (Metabolism and nutrition disorders) | 14 | 11 | 9
Diarrhea (Gastrointestinal disorders) | 10 | 11 | 12
Vomiting (Gastrointestinal disorders) | 12 | 11 | 9
White Blood Cell Decreased (Investigations) | 4 | 11 | 13
Weight Loss (Investigations) | 5 | 9 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 16
Infections And Infestations - Other, Pneumonia (Infections and infestations) | 10 | 9 | 5
Abdominal Pain (Gastrointestinal disorders) | 5 | 7 | 8
Thromboembolic Event (Vascular disorders) | 5 | 4 | 11
Proteinuria (Renal and urinary disorders) | 0 | 11 | 8
Rash (Skin and subcutaneous tissue disorders) | 6 | 8 | 5
Insomnia (Psychiatric disorders) | 9 | 5 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 9 | 4
Headache (Nervous system disorders) | 1 | 9 | 7
Hypertension (Vascular disorders) | 0 | 11 | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 2
Dizziness (Nervous system disorders) | 3 | 8 | 5
Mucositis (Gastrointestinal disorders) | 3 | 4 | 9
Non-Cardiac Chest Pain (General disorders) | 5 | 6 | 4
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 3 | 7
Fever (General disorders) | 10 | 3 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 | 5 | 5
Depression (Psychiatric disorders) | 5 | 6 | 2
Dysgeusia (Nervous system disorders) | 4 | 5 | 4
Urinary Tract Infection (Infections and infestations) | 2 | 5 | 6
Skin Infection (Infections and infestations) | 6 | 2 | 4
Anxiety (Psychiatric disorders) | 5 | 4 | 2
Confusion (Psychiatric disorders) | 2 | 4 | 5
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 7
Non-Cardiac Chest Pain (General disorders) | 5 | 5 | 1
Respiratory, Thoracic And Mediastinal Disorders - Other, Copd Exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 2
Sinusitis (Infections and infestations) | 0 | 4 | 5
Dysphagia (Gastrointestinal disorders) | 4 | 3 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 0 | 5
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1 | 4
Hypotension (Vascular disorders) | 3 | 0 | 5
Peripheral Sensory Neuropathy (Nervous system disorders) | 5 | 1 | 2
Oral Pain (Gastrointestinal disorders) | 1 | 5 | 2
Cardiac Disorders - Other, Tachycardia (Cardiac disorders) | 1 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites